CLINICAL TRIAL: NCT06496035
Title: Blood Flow Restriction Training Versus Traditional Rehab in Patients With Lower Extremity Fractures: Effect on Fracture Healing, Muscle Strength and Girth, and Return to Function
Brief Title: Blood Flow Restriction Training in Patients With Lower Extremity Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-0894
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Tibial Fractures; Lower Extremity Fracture
MeSH Terms: conditions — Tibial Fractures | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to experimental group performing exercise with blood flow restriction, or to the control group performing exercises without the device
Masking Description: Masking is not possible due to evident use or nonuse of device, and documentation in patient's chart.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blood flow restriction training (Experimental): Patients will perform exercises as directed by a Doctor of Physical Therapy with the use of blood flow restriction device
  Interventions: Device: Blood Flow Restriction with low load exercise
- Traditional physical therapy (Active Comparator): Patients perform physical therapy exercises guided by a Doctor of Physical Therapy without the use of a blood flow restriction device, as is current standard practice.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Device: Blood Flow Restriction with low load exercise — Cuff/tourniquet will be applied to proximal leg at hip crease and inflated to 60-80% of limb occlusion pressure to decrease venous blood flow in the limb while performing exercise.
  Arms: Blood flow restriction training
Other: Therapeutic Exercise — Exercise performed at appropriate load as guided by physical therapist
  Arms: Traditional physical therapy

SUMMARY:
This study will look at the effect of using a blood flow restriction device during low load strengthening exercises on patients with tibial shaft fractures, compared to patients performing exercise without the device. The study will compare muscle strength, muscle size, fracture healing, and return to normal function between the two groups.

DETAILED DESCRIPTION:
This study will examine the effect of blood flow restriction (BFR) training in patients with lower extremity fractures. Patients with tibial shaft fractures will be assigned to either the BFR group or control group. The BFR group will perform exercises with a blood flow restriction device, which occludes venous blood flow in the limb, while performing strengthening exercises as directed by a Doctor of Physical Therapy. The control group will perform the exercises without the device, as is current standard practice in physical therapy. Blood flow restriction training has been shown to prevent strength loss and muscle atrophy after surgery or injury, and studies suggest that it increases biomarkers of bone metabolism and tissue healing. The goal of this study is to examine the use of BFR in trauma patients using a defined protocol, and compare fracture healing, muscle strength, muscle girth, and subjective physical function between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult with closed tibial shaft fracture
* Ability to begin physical therapy treatment within 2 weeks post-operatively

Exclusion Criteria:

* History of osteoporosis or osteopenia
* Impaired circulation in the limb
* Active deep vein thrombosis
* Clotting disorders or other elevated risk of embolism
* Sickle cell anemia
* Infection in extremity
* Renal compromise
* Severe uncontrolled hypertension (SBP>180)
* Lymphedema
* Under age 18
* Pregnancy
* Prisoner

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Fracture healing | 6 weeks, 12 weeks, 6 months
  Tibial shaft fracture healing as measured by Radiographic Union Score for Tibial (RUST) fractures

SECONDARY OUTCOMES:
Muscle strength | 2 weeks, 4 weeks, 6 weeks, 12 weeks, and 6 months
  Knee extension and ankle plantarflexion strength measured with a dynamometer
Muscle girth | 2, 4, 6, 12 weeks and 6 months
  Quadriceps and gastrocnemius muscle girth measured 15 cm above and below joint line
Physical function | 2, 6,12 weeks and 6 months
  Subjective measure of function measured by Lower Extremity Functional Scale (LEFS)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Smith, PT, DPT, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No